CLINICAL TRIAL: NCT06293586
Title: A Comparison Between The Effects Of Peribulbar And Sub-tenon Blocks Combined With General Anesthesia On The Incidence Of Oculocardiac Reflex (OCR) During Pediatric Strabismus Surgery: A Double Blinded Randomised Control Study
Brief Title: Comparison Between Peribulbar And Sub-tenon Blocks on Oculocardiac Reflex (OCR) During Pediatric Strabismus Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Essam El-Din Zaki Bassyouni, assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MD-11-2022
Record Dates: First submitted 2024-02-20; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Anesthesia, Local; Ophthalmopathy; Strabismus; Pediatric ALL
Keywords: paracetamol; peribulbar block; sub-tenon block; pediatric strabismus surgery; oculocardiac reflex
MeSH Terms: conditions — Eye Diseases; Strabismus; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Peribulbar group (Group P) (Experimental): The peribulbar group (P group _ 40) received a peribulbar block with 0.25 mL/kg of a 1:1 local anesthetic mixture (LAM) of 0.5% bupivacaine and 2% lignocaine. Peribulbar block using a two-injection technique was performed by a second anesthetist under sterile conditions and before the application of surgical drapes. LAM was injected both infratemporal and superonasally using a 26-G needle, in contrast to the single infratemporal injection approach.
  Interventions: Procedure: peribulbar block
- sub-tenon group (group S) (Experimental): Children in the sub-Tenon group (sub-Tenon group (S), n _ 40) received a sub-Tenon block. Sub-Tenon's anesthesia was performed with 0.5% bupivacaine (0.08 ml/kg), bearing in mind not to exceed the maximum dose. Under sterile conditions, a 19- gauge curved blunt metallic cannula (25 mm) was inserted into sub-Tenon's space and the local anesthetic was injected by the ophthalmologist after the application of surgical drapes.
  Interventions: Procedure: sub-tenon block
- paracetamol (group C) (Active Comparator): Children in the paracetamol group received IV paracetamol (15 mg/kg) after induction of anesthesia before any surgical intervention.
  Interventions: Drug: Paracetamol

INTERVENTIONS:
Procedure: peribulbar block — Peribulbar block using a two-injection technique was performed by a second anesthetist under sterile conditions and before the application of surgical drapes. LAM was injected both infratemporal and superonasally using a 26-G needle, in contrast to the single infratemporal injection approach.
  Gentle digital oculopression was performed for 5 minutes
  Arms: Peribulbar group (Group P)
Procedure: sub-tenon block — Children in the sub-Tenon group received a sub-Tenon block. Sub-Tenon's anesthesia was performed with 0.5% bupivacaine (0.08 ml/kg), bearing in mind not to exceed the maximum dose. Under sterile conditions, a 19- gauge curved blunt metallic cannula (25 mm) was inserted into sub-Tenon's space and the local anesthetic was injected by the ophthalmologist after the application of surgical drapes.
  Arms: sub-tenon group (group S)
Drug: Paracetamol — Children in the control group received IV paracetamol (15 mg/kg) after induction of anesthesia before any surgical intervention.
  Other Names: paracetamol iv
  Arms: paracetamol (group C)

SUMMARY:
The aim of this study is to compare between peribulbar block and subtenon block as an adjunct to general anesthesia in children undergoing strabismus surgery on oculocardiac reflex (OCR), post-operative analgesia and postoperative vomiting. Both techniques will be compared to intra-operative intravenous (IV) paracetamol combined with general anesthesia as a sole anesthetic technique.

DETAILED DESCRIPTION:
120 children, American Society of Anaesthesiology (ASA) I or II, aged 6 to 13 years, scheduled for elective squint surgery under GA will be included in the study. Children with tumors or infections of the orbit, raised intraocular pressure, eye injury, airway abnormalities or who are blind in the eye other than that which will to be operated, will be excluded. Other exclusion criteria will include known allergy to local anaesthetics or nonsteroidal anti-inflammatory drugs (NSAIDS), steroid therapy, those with significant cardiac, respiratory, renal, hepatic, or neurological disorders, mentally challenged children, or parental refusal to participate.

All children will undergo a detailed preanesthetic evaluation including previous history of operations, drug history, physical examination (cardiovascular and respiratory systems, blood pressure, oxygen saturation, airway and dentition, body weight and height). During the pre-anesthesia evaluation, children will be encouraged to report postoperative pain, if present. All children will be fasted for a minimum of 4 hours and premedicated with oral midazolam 0.5 mg/kg 30 minutes before anaesthesia. Anesthesia will be induced with sevoflurane 6% in oxygen or intravenous (i.v.) propofol (2mg/kg), as appropriate for the child's age and preference. Following inhalational induction, an intravenous line will be placed. The airway will be secured using an appropriately sized endotracheal tube (ETT) following intravenous atracurium(0.5 mg.kg) and 1 to 3 min of mask ventilation using isoflurane 1.5% in oxygen.Anesthesia will then be maintained with isoflurane in air-oxygen and end tidal minimal alveolar concentration maintained at 1 to 1.3. ventilation will be established at 6-8ml per kg with a target PECO2 of 32 - 34 and will be adjusted accordingly.

Children will then be randomly allocated to one of three groups; by a nurse who will not participate in the study, reads the number contained in the envelope and makes group assignment.

Children in the control group (group C, n_20) will receive IV paracetamol (20mg/kg).

Children in the sub-tenon group (sub-tenon group (S), n _ 20) will receive a sub-tenon block. Sub-Tenon's anesthesia will be performed with 5% bupivacaine (0.08 ml/kg). Under sterile conditions, a 19-gauge curved, blunt metallic cannula (25 mm) will be inserted into sub-Tenon's space and the local anesthetic will be injected by the ophthalmologist.

The peribulbar group (P group _ 20) will receive peribulbar block with 0.25 mL/kg of a 1:1 mixture of 0.5% bupivacaine and 2% lignocaine containing hyaluronidase (500 IU hyaluronidase has been premixed with 30 mL 2% lignocaine). Peribulbar block using a two-injection technique will be performed by a second anaesthetist.

The children will not be aware to as which group they will be allocated into. Digital oculopression will be performed for 5 minutes. All blocks will be performed by one of the investigators. LAM will be injected both inferotemporallly and superonasally using a 26-G needle. Haemodynamic variables; electrocardiography (ECG), pulse oximetry, noninvasive blood pressure (NIBP) and end tidal carbon dioxide (PECO2); will be monitored continuously and Occurrence of oculocardiac reflex (OCR) will be recorded (either in the form of bradyarrhythmias mostly sinus bradycardia or o) . bradyarrhythmias which is the most common presentation of Oculocardiac reflex (OCR) will be considered as an acute decrease in heart rate below 60 beats/min and will be treated by asking the surgeon to stop stimulation and giving intravenous atropine (0.01 mg.kg), whereas other less common presentations of oculocardiac reflex (OCR) will be managed accordingly. All children will receive Dexamethasone (0.125mg/kg) 30 minutes before the end of surgery. At the end of the procedure, the ETT will be removed after reversing residual neuromuscular blockade with 50 μg·kg-1 neostigmine and 20 μg·kg-1 atropine and adequate spontaneous ventilation established.

Children will then be transferred to the recovery room, where they will be kept for 2 to 3 hours. On arrival in the recovery room, the child's' behavior and postoperative pain level will be assessed at 30 min by the recovery room nurse who will not be aware of the block using the modified objective pain scale (MOPS) [10] which assess pain via 5 points (crying, facial expressions, posture of the trunk, posture of the legs, and motor restlessness) with a minimum score of 0 and a maximum score of 10. 0-1 (no pain), 2-5 (mild), 6-7 (moderate), and 8-10 (severe) out of 10.

For pain judged as moderate or severe (MOPS > 5), ibuprofen 10mg/kg will be administered orally. After 2 hours in the recovery area, the children's pain will be assessed by Modified objective pain scale (MOPs) at 2 and 4 hours. Requirement of postoperative analgesia will be recorded. The incidence of PONV will be recorded. Numeric scoring will be used for PONV (0 = no nausea; 1 = nausea is present, but no vomiting; 3 = vomiting once within 30 min; 4 = vomiting two or more times within 30 min). Ondansetron (0.1 mg/kg, i.v.) will be given in cases of vomiting. The data collector will not be aware of the intervention the child will receive

ELIGIBILITY:
Inclusion Criteria:

* Participants were children (6-13 years), ASA I-II patients, scheduled to undergo strabismus surgery.

Exclusion Criteria:

* Children with tumors or infections of the orbit, raised intraocular pressure more than 20 mm Hg, axial length more than 28 mm, eye injury, airway abnormalities or who were blind in the eye other than that which was to be operated on were excluded. Other exclusion criteria included patients undergoing revision surgery, known allergy to local anesthetics or non-steroidal antiinflammatory drugs (NSAIDs), steroid therapy, parental refusal to participate and patients with INR more than 1.5 or with platelets less than 100.

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 140 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of intraoperative oculocardiac reflex (OCR) | 2 hours
  drop in heart rate below 60 bpm

SECONDARY OUTCOMES:
blood pressure | 2 hours
  blood pressure in mmhg will be recorded preop, after induction, and every 15 minutes.
heart rate | 2 hours
  heart rate as beats per minute will be recorded preop, after induction, and every 15 minutes.

OTHER OUTCOMES:
Post-operative pain using the MOPS | 4 hours
  pain assessed using the MOPS
Post-operative analgesia requirements | 4 hours
  pethidine 0.5 mg/kg was administered IV
The incidence of POV using numeric scoring | 2 hours
  using Numeric scoring at 30 minutes and 2h post-operative
Complications resulting from orbital regional anesthesia were recorded | 2 hours
  e.g.: subconjunctival hemorrhage, local anesthetic toxicity, chemosis, optic neuropathy, extra-ocular muscle paresis
Total intraoperative atropine requirements | 2 hours
  Brady arrhythmias intraoperatively which are the most common presentation of OCR was considered when an acute decrease in heart rate below 60 beats/min and was treated by asking the surgeon to stop stimulation and giving intravenous atropine (0.01 mg. kg)

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University faculty of medicine, Cairo, Egypt